CLINICAL TRIAL: NCT05905029
Title: Establishment of Biomechanical-based Rehabilitation Strategies for Pain-inducing Lifestyles in Degenerative Knee/Back Patients and for Artificial Intelligence-based Rehabilitation System
Brief Title: Establishment of Biomechanical- and AI- Based Rehabilitation Strategies for Pain Inducing Lifestyles
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principle investigator, Bundang CHA Hospital
Other Study IDs: 2022-11-015
Record Dates: First submitted 2023-05-29; First posted 2023-06-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Healthy; Degenerative Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To develop biomechanical indicators for pain-inducing lifestyles and apply lifestyle strategies for patients and confirm their effectiveness to be used in artificial intelligence-based digital treatment devices.

DETAILED DESCRIPTION:
To develop biomechanical indicators for pain-inducing lifestyles and apply lifestyle strategies for patients and confirm their effectiveness to be used in artificial intelligence-based digital treatment devices for patients who complain degenerative knee and back pain.

ELIGIBILITY:
1. Normal subjects

   * Inclusion criteria

     1. Over 19 years of age
     2. Those who scored '0' on the Knee/Back Pain Assessment Scale (VAS)
     3. After hearing a detailed explanation of this study and fully understanding it, the subject or legal representative voluntarily decides to participate and agrees in writing to observe the precautions
   * Exclusion criteria

     1. Patients who correspond to one or more of the following cannot participate in the study.
     2. Those with systemic infectious symptoms at the time of participation in the study
     3. Persons with poor systemic conditions such as unstable conditions of the cardiovascular system, digestive system, respiratory system, endocrine system, etc., and those with cerebrovascular disease
     4. Other cases where the researcher judges that participation in this study is not suitable (Patients who are participating in other studies or who have participated in other studies within the past 30 days can also participate in this study.)
2. Subjects who complain pain by degenrative changes in knee

   * Inclusion criteria

     1. Over 19 years of age
     2. Those who scored '1' or higher on the Knee Pain Assessment Scale (VAS)
     3. After hearing a detailed explanation of this study and fully understanding it, the subject or legal representative voluntarily decides to participate and agrees in writing to observe the precautions
   * Exclusion criteria

     1. Patients who correspond to one or more of the following cannot participate in the study.
     2. Those with systemic infectious symptoms at the time of participation in the study
     3. Persons with poor systemic conditions such as unstable conditions of the cardiovascular system, digestive system, respiratory system, endocrine system, etc., and those with cerebrovascular disease
     4. Other cases where the researcher judges that participation in this study is not suitable (Patients who are participating in other studies or who have participated in other studies within the past 30 days can also participate in this study.)
3. Subjects who complain pain by degenrative changes in back

   * Inclusion criteria

     1. Over 19 years of age
     2. Those with a back pain rating scale (VAS) of '1' or higher
     3. After hearing a detailed explanation of this study and fully understanding it, the subject or legal representative voluntarily decides to participate and agrees in writing to observe the precautions
   * Exclusion criteria

     1. Patients who correspond to one or more of the following cannot participate in the study.
     2. Those with systemic infectious symptoms at the time of participation in the study
     3. Persons with poor systemic conditions such as unstable conditions of the cardiovascular system, digestive system, respiratory system, endocrine system, etc., and those with cerebrovascular disease
     4. Other cases where the researcher judges that participation in this study is not suitable (Patients who are participating in other studies or who have participated in other studies within the past 30 days can also participate in this study.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and patients who complain pain by degenerative changes in knee or back
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Motion analysis | 1 day after screening assessment
  Motion capture analysis for kinetic and kinematic data

SECONDARY OUTCOMES:
Ground reaction force | 1 day after screening assessment
  GRF measurement for ground reaction force in newtone
EMG measurement | 1 day after screening assessment
  Electromyography in maximum voluntary contraction

CONTACTS AND LOCATIONS:
Overall Officials: Minyoung Kim, M.D., Ph.D., Principal Investigator — Bundang CHA Hospital
Locations (1):
- Department of Rehabilitation Medicine, CHA Bundang Medical Center, Seongnam, South Korea